CLINICAL TRIAL: NCT01967745
Title: Laparoscopic vs. Open Surgical Procedure in Management of Acute Appendicitis
Brief Title: Laparoscopic Versus Open Appendectomy
Status: Completed | Type: Observational
Sponsor: Varazdin General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 01091981
Record Dates: First submitted 2013-10-11; First posted 2013-10-23 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Acute Appendicitis
Keywords: open appendectomy; laparoscopic appendectomy; appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- laparoscopic appendectomy: The laparoscopic appendectomy was performed with three trocars, placed in the periumbilical area, right midabdomen, and forceps.
  Interventions: Procedure: laparoscopic appendectomy
- open appendectomy: The open appendectomy was carried out in the standard way with McBurney muscle splitting incision (in supine position).
  Interventions: Procedure: open appendectomy

INTERVENTIONS:
Procedure: laparoscopic appendectomy — The laparoscopic appendectomy was performed with three trocars. Pneumoperitoneum was created using an open Hasson technique. The mesoappendix was divided using a harmonic scalpel or endoscopic tissue fusion device. The appendix was divided by placing one endoscopic loop and cut with harmonic scalpel. The specimen was removed through the umbilical port.
  Other Names: harmonic scalpel (UltraCision Ethicon ®); fusion device (Covidien LigaSure™); stapling device (Covidien Endo GIA™)
  Groups: laparoscopic appendectomy
Procedure: open appendectomy — The open appendectomy was carried out in the standard way with McBurney muscle splitting incision (in supine position).
  Groups: open appendectomy

SUMMARY:
Comparison of open and laparoscopic appendectomy

DETAILED DESCRIPTION:
Adult patients with presumptive diagnosis of acute appendicitis were were operated by laparoscopic appendectomy or open appendectomy group during a three-year period (between 2007 and 2009).

ELIGIBILITY:
Inclusion Criteria:

* patients older than 16 years with presumptive diagnosis of acute appendicitis

Exclusion Criteria:Appendectomy performed during diagnostic laparoscopy and incidental appendectomies patients with:

* cirrhosis
* ascites
* coagulation disorder
* diffuse peritonitis
* shock on admission
* large ventral hernia. Appendectomy performed during diagnostic laparoscopy and incidental appendectomies were also excluded

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with clinical, laboratory, and radiologic signs of acute appendicitis
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Cost of hospitalization based on the final hospital bills | from the beginning of the surgery till discharge from hospital (an expected average of 8 days, maximmum 20 days)

SECONDARY OUTCOMES:
Analgesia demands | from the beginning of the surgery till discharge from hospital (an expected average of 8 days, maximmum 20 days)
  The number of doses of analgesics, and time from surgery to the last dose of analgesics.
Complications | during first 4 weeks after the surgery
  No. of wound infection and intrabdominal abscesses.
Length of hospital stay | from the beginning of the surgery till discharge from hospital (an expected average of 8 days, maximmum 20 days)
  No. of days from surgery to discharge of hospital
Time until resumption of clear liquid and regular diet | from the beginning of the surgery to the resumption (an expected average 2 days after the surgery)
  No. of days from surgery to the resumption of clear liquid and regular diet

CONTACTS AND LOCATIONS:
Overall Officials: Ranko Stare, MD, PhD, Principal Investigator — Varazdin General Hospital
Locations (1):
- Varazdin General Hospital, Varaždin, Croatia